CLINICAL TRIAL: NCT00980785
Title: Studying the Effects of Antihypertensives on Individuals at Risk for Alzheimer's
Acronym: SEAIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-1353; H-2009-0036 (Other: UW Madison IRB); A534255 (Other: UW, Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW, Madison)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease; Hypertension
Keywords: Alzheimer's Disease; Hypertension
MeSH Terms: conditions — Alzheimer Disease; Hypertension | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo
- Active (Experimental): Ramipril 5mg/day
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — Ramipril 5 mg/day
  Other Names: Altace
  Arms: Active
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Angiotensin converting enzyme inhibitors (ACE-I) are a group of blood pressure-lowering medicines. Some studies suggest that ACE-I, such as ramipril, may help prevent Alzheimer's disease (AD). The purpose of the research is to see how ramipril affects a substance in the body called beta-amyloid. Beta-amyloid is found in the brain and in the liquid around the brain and spinal cord. High amounts of beta-amyloid may be associated with a greater risk of getting Alzheimer's disease. This study will see if ramipril can lower the amount of beta-amyloid in the spinal fluid. This study will also see if ramipril affects blood vessel function and memory and thinking. The investigators hope that future studies will show whether ramipril might prevent memory loss and decrease the chance of developing Alzheimer's disease.

DETAILED DESCRIPTION:
High blood pressure (BP) in midlife is predictive of Alzheimer's disease (AD) in later life. Similarly, reductions in BP are associated with protection against AD. Treatment with antihypertensive medications, specifically angiotensin converting enzyme inhibitors (ACE-I) such as ramipril, is associated with up to a 55% reduction in the prevalence of AD, suggesting a potentially promising role for ACE-I in the prevention of AD. It is unknown however 1) whether ACE-Is will have the same effect on Cerebrospinal fluid (CSF) Aβ levels in humans as in animal models 2) whether ACE-Is induce changes associated with vascular function (i.e. levels of CSF angiotensin converting enzyme (ACE) and peripheral endothelial function) and 3) whether there are interactions between ACE-I-induced changes in CSF Aβ, CSF ACE and indices of vascular function.

One mechanism by which antihypertensives may protect against AD is via Aβ neuropathology. In order to better understand the mechanisms through which ACE-I may modify CSF Aβ and possibly AD risk, we propose a randomized, double-blind, placebo-controlled pilot clinical trial, enrolling 20 middle-aged (age range 40 - 65 years), mildly hypertensive (between 130 - 160 mmHg mean systolic and between 85 - 100 mmHg mean diastolic) participants, who are adult children of an individual with AD. The main objective of this trial is to examine the effects of the ACE-I, ramipril, on 1) CSF Aβ levels 2) CSF ACE levels and 3) peripheral endothelial function as measured by brachial artery flow-mediated vasodilation (FMD) and aortic augmentation index (AAIx), in middle-aged adults with mildly elevated BP, who are at increased risk of developing AD.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40 and 65
* Mean resting blood pressure between 130-160 systolic and 85-100 diastolic
* Parent with Alzheimer's Disease

Exclusion Criteria:

* Current involvement in another investigational drug trial.
* Potassium > 5.0
* Dementia based on DSMIV criteria
* Mini-Mental State Exam (MMSE) score < 27
* Current blood pressure medication (< 4 months from screening)
* Weight loss medication
* Contraindications for LP
* Know diagnosis or history of hospitalization due to congestive heart failure
* Elevated creatinine (females > 1.3 mg/dL or males > 1.4 mg/dL at baseline)
* Diabetes Type I and II
* Know adverse reaction to an ACE-I or an angiotensin receptor blocker
* Pregnant of nursing women

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04-09 (Actual); Primary Completion 2011-07-26 (Actual); Study Completion 2011-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Carlsson, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconisn Alzheimer's Disease Research Center, Madison, Wisconsin, United States

REFERENCES:
- [Background] Wharton W, Stein JH, Korcarz C, Sachs J, Olson SR, Zetterberg H, Dowling M, Ye S, Gleason CE, Underbakke G, Jacobson LE, Johnson SC, Sager MA, Asthana S, Carlsson CM. The effects of ramipril in individuals at risk for Alzheimer's disease: results of a pilot clinical trial. J Alzheimers Dis. 2012;32(1):147-56. doi: 10.3233/JAD-2012-120763. PMID 22776970
- See also: Related Info — http://wisconsinadrc.wisc.edu/prevention_research.shtml
- See also: The Effects of Ramipril in Individuals at Risk for Alzheimer's Disease: Results of a Pilot Clinical Trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3593582/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Wisconsin Alzheimer's Disease Research Center (ADRC) registry and from the community for the clinical trial, Studying the Effects of Antihypertensives in Individuals at Risk for Alzheimer's (SEAIRA).
Period: Overall Study
Arm/Group | Placebo | Active
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (6.7) | 56.3 (6.1) | 54.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebrospinal Fluid (CSF) Amyloid Beta-42 (Aβ42) Levels Between Baseline and Month 4 in Subjects Taking Ramipril vs Subjects on Placebo
Description: CSF Aβ42 levels will be measured from the cerebrospinal fluid taken from subjects on ramipril or placebo at the baseline visit and month 4 and will be measured by Dr. Henrik Zetterberg's laboratory.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | Active
Number analyzed (Participants) | 6 | 8
pg/ml | -22.5 (78.7) | -31.71 (90.6)
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Mann-Whitney test; p = 0.836, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -22.5, Standard Deviation 78.7
Statistical Analysis 2: Comparison: Active; Test type: Other — Mann-Whitney Test; p = 0.836, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -31.71, Standard Deviation 90.6

2. Secondary Outcome: Change in CSF Angiotensin Converting Enzyme (ACE) Levels Between Baseline and Month 4 in Subjects Taking Ramipril vs Subjects on Placebo
Description: CSF ACE levels will be measured from the cerebrospinal fluid taken from subjects on Ramipril or placebo at the baseline visit and month 4 and will be measured by ARUP® laboratories by spectrophotometric enzymatic assay.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Active
Number analyzed (Participants) | 6 | 8
U/L | -0.10 (0.21) | -0.63 (0.32)
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Mann-Whitney Test; p = 0.009, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.10, Standard Deviation 0.21
Statistical Analysis 2: Comparison: Active; Test type: Other — Mann-Whitney Test; p = 0.009, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.63, Standard Deviation 0.32

3. Secondary Outcome: Change in Flow-mediated Vasodilation (FMD) Between Baseline and Month 4 in Subjects Taking Ramipril vs Subjects on Placebo
Description: FMD is calculated as the ratio of brachial artery diameter after reactive hyperemia to baseline diameter, expressed as percentage change. FMD for each subject (ramipril v placebo) will be measured at baseline and month 4, observing any differences.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Active
Number analyzed (Participants) | 6 | 8
Percentage change | -0.70 (1.56) | -0.29 (1.23)
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Mann-Whitney Test; p = 0.755, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.70, Standard Deviation 1.56
Statistical Analysis 2: Comparison: Active; Test type: Other — Mann-Whitney test; p = 0.755, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.29, Standard Deviation 1.23

4. Secondary Outcome: Change in Augmentation Index (%) Between Baseline and Month 4 in Subjects Taking Ramipril vs Subjects on Placebo
Description: Pulse wave velocity was measured using an AtCor SphymoCor Px tonometry system. A small pressure transducer was placed on the skin at the point the arterial pulsation of the right common carotid and right radial arteries. A Millar micromanometer is in the tip of the probe. Using a generalized transfer function, the distance between these pressure points, and the peripheral arterial waveforms, a central aortic pressure signal is derived, from which aortic augmentation index is determined.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Active
Number analyzed (Participants) | 6 | 8
Percentage change | 1.7 (8.9) | -1.8 (2.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Other — Mann-Whitney test; p = 0.491, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.7, Standard Deviation 8.9
Statistical Analysis 2: Comparison: Active; Test type: Other — Mann-Whitney test; p = 0.491, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.8, Standard Deviation 2.2

ADVERSE EVENTS:
Arm/Group | Placebo | Active
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

LIMITATIONS AND CAVEATS:
Limitations included small sample size, short duration of trial, and lack of A-beta neuropathology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT00980785/Prot_SAP_000.pdf